CLINICAL TRIAL: NCT05252884
Title: Comparison of Routine Prophylactic Calcium + Calcitriol and Selective Use Based on PTH for the Prevention of Postoperative Hypocalcemia in Patients With Total Thyroidectomy. Randomized Clinical Trial
Brief Title: Calcium+Calcitriol Versus PTH for the Prevention of Hypocalcemia in Thyroidectomy. Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Excelencia en Enfermedades de Cabeza y Cuello (Other)
Collaborators: IPS universitaria (Unknown); Hospital San Vicente Fundación (Other); Clinica Las Vegas- Grupo QuironSalud (Unknown)
Responsible Party: Principal Investigator, Alvaro Sanabria, Scientific Director, Centro de Excelencia en Enfermedades de Cabeza y Cuello
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Cancer; Goiter; Thyroiditis; Hyperthyroidism
Keywords: thyroidectomy, hypocalcemia, randomized clinical trial
MeSH Terms: conditions — Thyroid Neoplasms; Goiter; Thyroiditis; Hyperthyroidism; Hypocalcemia | interventions — Calcitriol; Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, multicenter stratified clinical trial with 1:1 allocation.
Who Masked: Participant, Care Provider
Masking Description: It will be randomized by the block method and will be stratified by institution, type of disease (benign vs. malignant) and presence or absence of central voiding. This will be done centrally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium correction according to PTH levels (Experimental): A PTH blood test will be performed 4 hours post-thyroidectomy.
  Interventions: Diagnostic Test: calcium correction according to PTH levels
- routine postoperative calcium and calcitriol (Active Comparator): The patient will receive Calcium carbonate + calcitriol
  Interventions: Drug: routine postoperative calcium and calcitriol

INTERVENTIONS:
Diagnostic Test: calcium correction according to PTH levels — A PTH blood test will be performed 4 hours post-thyroidectomy. If the PTH result is >15 pg/mL, the patient will be discharged without calcium intake; if PTH < 15 pg/mL, start a dose of 1200 mg Calcium carbonate every 8 hours + 0.25 mcg of calcitriol every 12 hours orally for 15 days
  Other Names: PTH
  Arms: calcium correction according to PTH levels
Drug: routine postoperative calcium and calcitriol — The patient will receive a dose of 1,200 mg Calcium carbonate every 8 hours + 0.25 mcg of calcitriol every 12 hours orally for 15 days, starting on the same day as the intervention.
  Other Names: calcium carbonate, calcitriol
  Arms: routine postoperative calcium and calcitriol

SUMMARY:
The objective of this study is to compare the frequency of post-thyroidectomy symptomatic and biochemical hypocalcaemia between the strategy of routine prophylactic calcium + calcitriol vs the administration of calcium guided by PTH values.

DETAILED DESCRIPTION:
Postoperative hypocalcaemia is the most common complication that occurs in patients undergoing total thyroidectomy 1, with a frequency between 15 and 30%. 1-3 In the vast majority of cases, this complication is transitory, and only 1-3% manifest definitively. 4.5 Hypocalcemia is produced by surgical manipulation of the parathyroid glands, where their vascularization may be compromised, by stunning, or by inadvertent removal of the glands during thyroidectomy. 3,4 Other risk factors that have been associated include bilateral resection, inflammatory disease, and parathyroid reimplantation.1,6 Despite minimal manipulation during the surgical procedure, episodes of postoperative hypocalcemia continue to occur. To reduce the frequency of appearance and obtain symptomatic relief in the patient, several preventive strategies have been developed, 4,7-9 among which are the postoperative prophylactic administration of calcium + calcitriol 5,9 and the postoperative measurement of parathyroid hormone ( PTH) as a reference for oral calcium administration. 4,10 These strategies differ in the frequency of adverse events and cost. To date, these two interventions have not been directly compared in a clinical trial to determine which of them offers greater effectiveness and fewer adverse events and costs, and their use is made according to the individual preferences of the surgeon. A randomized clinical trial would offer information of high methodological quality for the standardization of conduct.

Research Question In a postoperative total thyroidectomy patient, is the calcium + calcitriol administration strategy based on postoperative PTH measurement superior to the routine prophylactic administration of calcium + calcitriol to reduce the frequency of symptomatic and postoperative biochemical hypocalcaemia?

Justification Postoperative hypocalcaemia is a condition that occurs in up to a third of postoperative total thyroidectomy patients. Hypocalcaemia worsens the clinical condition of the patient, implies prolongations of the hospital stay, readmissions and use of medications. 2,3,6 In addition to an adequate surgical technique, its prevention involves pharmacological interventions and diagnostic tests.

Among the alternatives currently used is the prophylactic administration of calcium and calcitriol for two weeks. 11 Despite being a cheap and safe strategy, it has uncomfortable side effects for the patient such as constipation, epigastric pain, metallic taste, loss of appetite and mood changes. 12,13 Due to this, several authors have proposed the measurement of calcium or PTH in the immediate postoperative period as a reference to decide the need for oral administration of calcium and calcitriol, thus avoiding unnecessary use in patients with normal values. 2,4,8,10,11 Theoretically, a measurement of PTH >10 pg/ml in the postoperative period would allow predicting patients who are at greater risk of developing hypocalcaemia than those who are not and can be discharged without taking calcium + calcitriol, but studies are very heterogeneous and difficult to compare with each other. 2.14 Recently, a meta-analysis evaluated the strategy of administration of calcium + calcitriol vs calcium measurement with advantages for the first 10, but there are few clinical trials that compare this strategy with postoperative PTH measurement. 14 Because this surgical group performs outpatient management after thyroidectomy, defining which of the two strategies offers greater effectiveness and a better profile of adverse events is of the utmost importance, as it would allow making general recommendations and adjusting current institutional protocols. On the other hand, the result of this trial would be a potential source of information to evaluate the cost-effectiveness of interventions in the future.

Aim: To compare the frequency of post-thyroidectomy symptomatic and biochemical hypocalcaemia between the strategy of routine prophylactic calcium + calcitriol vs the administration of calcium guided by PTH values.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing total thyroidectomy who meet the following criteria: Patients over 18 years of age, Benign (goiter, thyroiditis, hyperthyroidism) or malignant (carcinoma) diagnosis, Patients who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

- Patients with parathyroid surgery in conjunction with thyroidectomy, Patients with prior parathyroid disease for other causes (hyperparathyroidism primary or secondary to kidney disease, etc.), Patients with anaplastic carcinoma or lymphoma, Patients undergoing total thyroidectomy for causes other than thyroid disease such as, for example, total laryngectomy or pharyngo-laryngectomy that, due to margins or direct extension, require thyroidectomy. , Altered cognitive state that interfered or made the evaluation impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
symptomatic hypocalcaemia | 15 days
  The presence of symptomatic hypocalcaemia in the postoperative period of thyroidectomy defined according to the scale proposed by Wilde et al. (hypoparathyroid patient questionnaire HPQ) Min value 0 Max value 60 Higher scores represent worst symptoms

SECONDARY OUTCOMES:
Biochemical hypocalcemia | 48 hours and 15 days postoperatively
  Biochemical hypocalcemia defined as serum calcium < 8 mg/dL or PTH < 15
Adverse events of the medication | 15 days
  Adverse events of the medication (calcium+calcitriol) included in the scale of Wilde et al.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Sanabria, MD, Principal Investigator — Centro de Excelencia en Enfermedades de Cabeza y Cuello
Locations (2):
- Colombia (2):
  - Hospital Alma Mater de Antioquia, Medellín, Antioquia
  - Hospital Universitario San Vicente Fundacion, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abboud B, Sargi Z, Akkam M, Sleilaty F. Risk factors for postthyroidectomy hypocalcemia. J Am Coll Surg. 2002 Oct;195(4):456-61. doi: 10.1016/s1072-7515(02)01310-8. PMID 12375749
- [Background] Mathur A, Nagarajan N, Kahan S, Schneider EB, Zeiger MA. Association of Parathyroid Hormone Level With Postthyroidectomy Hypocalcemia: A Systematic Review. JAMA Surg. 2018 Jan 1;153(1):69-76. doi: 10.1001/jamasurg.2017.3398. PMID 29167863
- [Background] Terris DJ, Snyder S, Carneiro-Pla D, Inabnet WB 3rd, Kandil E, Orloff L, Shindo M, Tufano RP, Tuttle RM, Urken M, Yeh MW; American Thyroid Association Surgical Affairs Committee Writing Task Force. American Thyroid Association statement on outpatient thyroidectomy. Thyroid. 2013 Oct;23(10):1193-202. doi: 10.1089/thy.2013.0049. Epub 2013 Sep 14. PMID 23742254
- [Background] Dedivitis RA, Aires FT, Cernea CR. Hypoparathyroidism after thyroidectomy: prevention, assessment and management. Curr Opin Otolaryngol Head Neck Surg. 2017 Apr;25(2):142-146. doi: 10.1097/MOO.0000000000000346. PMID 28267706
- [Background] Sanabria A, Dominguez LC, Vega V, Osorio C, Duarte D. Routine postoperative administration of vitamin D and calcium after total thyroidectomy: a meta-analysis. Int J Surg. 2011;9(1):46-51. doi: 10.1016/j.ijsu.2010.08.006. Epub 2010 Sep 8. PMID 20804871
- [Background] Iglesias P, Diez JJ. Endocrine Complications of Surgical Treatment of Thyroid Cancer: An Update. Exp Clin Endocrinol Diabetes. 2017 Sep;125(8):497-505. doi: 10.1055/s-0043-106441. Epub 2017 Apr 25. PMID 28444664
- [Background] Leoncini E, Ricciardi W, Cadoni G, Arzani D, Petrelli L, Paludetti G, Brennan P, Luce D, Stucker I, Matsuo K, Talamini R, La Vecchia C, Olshan AF, Winn DM, Herrero R, Franceschi S, Castellsague X, Muscat J, Morgenstern H, Zhang ZF, Levi F, Dal Maso L, Kelsey K, McClean M, Vaughan TL, Lazarus P, Purdue MP, Hayes RB, Chen C, Schwartz SM, Shangina O, Koifman S, Ahrens W, Matos E, Lagiou P, Lissowska J, Szeszenia-Dabrowska N, Fernandez L, Menezes A, Agudo A, Daudt AW, Richiardi L, Kjaerheim K, Mates D, Betka J, Yu GP, Schantz S, Simonato L, Brenner H, Conway DI, Macfarlane TV, Thomson P, Fabianova E, Znaor A, Rudnai P, Healy C, Boffetta P, Chuang SC, Lee YC, Hashibe M, Boccia S. Adult height and head and neck cancer: a pooled analysis within the INHANCE Consortium. Eur J Epidemiol. 2014 Jan;29(1):35-48. doi: 10.1007/s10654-013-9863-2. Epub 2013 Nov 24. PMID 24271556
- [Background] Carr AA, Yen TW, Fareau GG, Cayo AK, Misustin SM, Evans DB, Wang TS. A single parathyroid hormone level obtained 4 hours after total thyroidectomy predicts the need for postoperative calcium supplementation. J Am Coll Surg. 2014 Oct;219(4):757-64. doi: 10.1016/j.jamcollsurg.2014.06.003. Epub 2014 Jun 18. PMID 25053220
- [Background] Arer IM, Kus M, Akkapulu N, Aytac HO, Yabanoglu H, Caliskan K, Tarim MA. Prophylactic oral calcium supplementation therapy to prevent early post thyroidectomy hypocalcemia and evaluation of postoperative parathyroid hormone levels to detect hypocalcemia: A prospective randomized study. Int J Surg. 2017 Feb;38:9-14. doi: 10.1016/j.ijsu.2016.12.041. Epub 2016 Dec 27. PMID 28039060
- [Background] Sanabria A, Rojas A, Arevalo J. Meta-analysis of routine calcium/vitamin D3 supplementation versus serum calcium level-based strategy to prevent postoperative hypocalcaemia after thyroidectomy. Br J Surg. 2019 Aug;106(9):1126-1137. doi: 10.1002/bjs.11216. Epub 2019 Jun 25. PMID 31236917
- [Background] Cayo AK, Yen TW, Misustin SM, Wall K, Wilson SD, Evans DB, Wang TS. Predicting the need for calcium and calcitriol supplementation after total thyroidectomy: results of a prospective, randomized study. Surgery. 2012 Dec;152(6):1059-67. doi: 10.1016/j.surg.2012.08.030. Epub 2012 Oct 13. PMID 23068088
- [Background] Harvey NC, Biver E, Kaufman JM, Bauer J, Branco J, Brandi ML, Bruyere O, Coxam V, Cruz-Jentoft A, Czerwinski E, Dimai H, Fardellone P, Landi F, Reginster JY, Dawson-Hughes B, Kanis JA, Rizzoli R, Cooper C. The role of calcium supplementation in healthy musculoskeletal ageing : An expert consensus meeting of the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO) and the International Foundation for Osteoporosis (IOF). Osteoporos Int. 2017 Feb;28(2):447-462. doi: 10.1007/s00198-016-3773-6. Epub 2016 Oct 20. PMID 27761590
- [Background] Sanaei M, Banasiri M, Shafiee G, Rostami M, Alizad S, Ebrahimi M, Larijani B, Heshmat R. Calcium vitamin D3 supplementation in clinical practice: side effect and satisfaction. J Diabetes Metab Disord. 2016 Mar 29;15:9. doi: 10.1186/s40200-016-0231-0. eCollection 2015. PMID 27030820
- [Background] Houlton JJ, Pechter W, Steward DL. PACU PTH facilitates safe outpatient total thyroidectomy. Otolaryngol Head Neck Surg. 2011 Jan;144(1):43-7. doi: 10.1177/0194599810390453. PMID 21493385